CLINICAL TRIAL: NCT03737422
Title: Evaluation of the Effects of Hesperidin and Flaxseed Supplementation in Patients With Prediabetes
Brief Title: The Effects of Hesperidin and Flaxseed in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6781
Record Dates: First submitted 2018-10-11; First posted 2018-11-09 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2018-11

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Hesperidin; Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hesperidin and flaxseed (Active Comparator)
  Interventions: Dietary Supplement: hesperidin and flaxseed
- control (Placebo Comparator)
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: hesperidin and flaxseed — 2 capsuls hesperidin and 30 g flaxseed
  Arms: hesperidin and flaxseed
Other: control — no supplementation
  Arms: control

SUMMARY:
To study the effects of Hesperidin and flaxseed supplement in patients with prediabetes, 50 patients will be randomly allocated to control group or 2 capsules Hesperidin and 30 gram flaxseed for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, lipid profiles, blood pressure, blood sugar, inflammatory and anthropometric factors will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years prediabetes: impaired fasting glucose (>100 mg/dL) and/or HbA1C 5.7% to 6.5%, and overweight or obese with body mass index range of 25 to 40 kg/m2

Exclusion Criteria:

* pregnancy or lactation
* A history of Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* Following program to lose weight in recent 3 mo

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
prediabetes | 12 weeks
  number of participants with normal plasma glucose

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

REFERENCES:
- [Derived] Yari Z, Naser-Nakhaee Z, Karimi-Shahrbabak E, Cheraghpour M, Hedayati M, Mohaghegh SM, Ommi S, Hekmatdoost A. Combination therapy of flaxseed and hesperidin enhances the effectiveness of lifestyle modification in cardiovascular risk control in prediabetes: a randomized controlled trial. Diabetol Metab Syndr. 2021 Jan 6;13(1):3. doi: 10.1186/s13098-020-00619-y. PMID 33402222